CLINICAL TRIAL: NCT00316121
Title: A Prospective, Multicenter, Randomized Study Comparing the Use of HEALOS® to Autograft in a Transforaminal Lumbar Interbody Fusion (TLIF) Approach
Brief Title: Safety and Efficacy Study of Healos as a Bone Replacement to Treat Degenerative Disc Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanced Technologies and Regenerative Medicine, LLC (ATRM) (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Manny Lazaro, MS, Advanced Technologies and Regenerative Medicine, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-HEALOS-01
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Degenerative Disc Disease
Keywords: One or Two Level Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

ARMS (2):
- 1 (Experimental)
  Interventions: Device: HEALOS and Leopard Cage
- 2 (Active Comparator)
  Interventions: Device: Leopard Cage and Autograft

INTERVENTIONS:
Device: HEALOS and Leopard Cage — Placement in interbody space
  Arms: 1
Device: Leopard Cage and Autograft — Placement in the interbody space
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of HEALOS compared with autograft using the transforaminal lumbar interbody fusion (TLIF) method.

ELIGIBILITY:
Inclusion Criteria:

* Persistent back and/or leg pain refractory to 6 months of non-surgical therapy
* Male or female 18 to 70 years of age (inclusive)
* Objective evidence of significant disc degeneration at one or two adjacent lumbar level(s) from L2/L3 to L5/S1

Exclusion Criteria:

* Significant disc degeneration at more than two adjacent levels
* Greater than Grade II spondylolisthesis
* Prior fusion surgery of the lumbar spine (prior discectomies and intradiscal electrothermal therapy [IDET] are allowed)
* Insulin-dependent diabetes mellitus
* Pregnant or lactating, or wishes to become pregnant within the 24 month duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Brandon, Florida
  - Jacksonville, Florida
  - Savannah, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Annapolis, Maryland
  - Billings, Montana
  - Williamsville, New York
  - Norwood, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Temple, Texas
  - Salt Lake City, Utah
  - Spokane, Washington
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 3Apr06 to 31Dec07. Subjects were seen at medical clinics/hospitals, usually by their regular doctor and not found through ads. Subjects were asked to enroll if they were having back surgery for back pain. Enrollment was stopped for administrative reasons at 138 subjects; the per protocol plan was at least 350 subjects.
Pre-assignment Details: 220 subjects were screened and 82 were excluded (59 did not meet criteria and 23 refused participation).Use of non-steroidal anti-inflammatory medications or cyclooxygenase-II (COX-2) inhibitors (a non-steroidal anti-inflammatory drug that directly targets COX-2, an enzyme responsible for inflammation and pain) at time of surgery were exclusionary.
Groups:
- HEALOS: HEALOS is a synthetic bone graft material made of collagen (a fibrous protein) and hydroxyapatite (a natural mineral structure). The collagen is a bovine derivative (obtained from cows). HEALOS is similar to what is found in natural bone and has the clearance of the U.S. Food and Drug Administration for use in filling bony voids or gaps of the skeletal system. It is combined with bone marrow (a vascular or vessel-like tissue found in the cavity of bone) to form new bone. HEALOS with bone marrow aspirate is currently available for use in a procedure where rods and screws are placed in the back with graft material to fuse the vertebrae.
  The Leopard cage is a spinal implant made of a material called carbon fiber. HEALOS, when used with the Leopard Cage is an investigational device. An investigational device is one that is being tested and has not yet received approval from the Food and Drug Administration for the use in which it is being tested.
- Control: Autograft is bone taken from the subject's own hip and placed in and around the spinal implant and spinal instrumentation. Local bone (bone from the area of surgery and placed in the fusion site) may be used in combination with autograft.
Period: Overall Study
Arm/Group | HEALOS | Control
Started | 92 | 46
Completed | 70 | 37
Not Completed | 22 | 9
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 14 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Reason is missing | 1 | 0
Not completed — Subject relocated | 1 | 1
Not completed — Subject refused to return | 1 | 0
Not completed — Subject no show for visit x 3 | 1 | 0
Not completed — Subject did not have 24 month visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEALOS | Control | Total
Number analyzed (Participants) | 92 | 46 | 138
Age Continuous [Mean (Full Range); unit: Years] — Between 18-70 years old
  Years | 47.4 [21 to 68] | 49.5 [22 to 70] | 48.45 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 27 | 84
  Male | 35 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Subject Success (Success is Defined Only if All of These Criteria Are Fulfilled)
Description: Success is bridging bone, slip of study level versus adjacent levels less than 3 millimeters, angulation less than 5 degrees, 15 point increase in Oswestry Disability Index (ODI) (how back/leg trouble affects activities of daily living), no new problems in motor strength in legs, presence/absence of pain on leg raise, sensation intact on thigh/leg/foot reflexes of the knees/ankles, no permanent/serious complications, no revision/removal/reoperation/supplemental fixation. The ODI is on a 6 point scale from 0 (no pain/no impact on duties) to 5 (worst pain ever/unable to perform duties).
Time Frame: 24 months
Population: Safety Population:All subjects treated. Full Analysis Set(FAS):Subset of Safety Pop. w/follow up. All effectiveness measures were to be assessed on FAS. FAS is intent-to-treat pop. Per Protocol: Subset of FAS who complete study, treated as randomized w/no major protocol deviations. All analyses were to be on this subset.
Measure: Number; unit: Subjects
Arm/Group | HEALOS | Control
Number analyzed (Participants) | 71 | 39
Subjects | 0 [0.0 to 5.1] | 0 [0.0 to 9.0]

ADVERSE EVENTS:
Time Frame: 4 years and 7 months
Description: Regular assessments made via study visits.
Arm/Group | HEALOS | Control
Serious Adverse Events (participants affected / at risk) | 23/92 | 13/46
Other Adverse Events (participants affected / at risk) | 77/92 | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEALOS (N=92) | Control (N=46)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalization
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalization
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) — 2 hospitalizations for the same patient
Implant Site Pain (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Hospitalization
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Hospitalization after a fall
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) — Hospitalization x4
Intervertebral Discitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) — Hospitalization x6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Hospitalization x2
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 1 (1) | 0 (0) — Hospitalization
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Cystocele (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEALOS (N=92) | Control (N=46)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) — Does not meet the criteria for seriousness
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 10 (10) | 8 (10) — Does not meet the criteria for seriousness
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) — Does not meet the criteria for seriousness
Asthenia (General disorders) | 4 (5) | 5 (5)
Chest Pain (General disorders) | 6 (7) | 1 (1)
Oedema Peripheral (General disorders) | 3 (3) | 5 (8)
Pain (General disorders) | 1 (1) | 3 (4)
Pyrexia (General disorders) | 8 (8) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 4 (6) — Does not meet criteria for seriousness
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Back Injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 8 (10)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
Road Traffic Accident (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (16) | 8 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 30 (34) | 21 (28) — Does not meet criteria for seriousness
Bursitis (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) — Does not meet criteria for seriousness
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) — Does not meet criteria for seriousness
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 14 (23) — Does not meet criteria for seriousness
Cervicobrachial Syndrome (Nervous system disorders) | 6 (7) | 0 (0) — Does not meet criteria for seriousness
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 8 (11) | 8 (12)
Hyporeflexia (Nervous system disorders) | 3 (3) | 4 (7)
Paraesthesia (Nervous system disorders) | 11 (15) | 4 (4)
Sensory Loss (Nervous system disorders) | 8 (9) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 7 (7) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Stringent criteria for endpoint.Minimum sample size not reached; no hypothesis testing.High portion of current/prior smokers in both groups may impact fusion success.Product usage was appropriate and not low.This study is not on label for HEALOS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot publish the results without consent of Sponsor. The results must be given to Sponsor 60 days prior to use. This review is not meant to curtail distribution of data, but to identify confidential material and/or to review the content for conformance to regulations. The Sponsor has the right to edit materials to preserve confidentiality of proprietary information. If requested, the Institution and PI will withhold publication for 60 days to allow for filing of a patent application.